CLINICAL TRIAL: NCT07188844
Title: An Open-Label Extension Study to Assess Long-term Safety and Tolerability of Batoclimab in Adult Participants With Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
Brief Title: An Open-Label Extension Study of Batoclimab in Adult Participants With Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Immunovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMVT-1401-2402
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy
Keywords: Chronic Inflammatory Demyelinating Polyneuropathy; IMVT-1401; Monoclonal antibody; Autoimmune disorders; Batoclimab
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Batoclimab (Experimental)
  Interventions: Drug: Batoclimab

INTERVENTIONS:
Drug: Batoclimab — Batoclimab 340 mg SC QW
  Other Names: IMVT-1401

SUMMARY:
This is an open-label extension (OLE) study designed to evaluate the long-term safety and tolerability of batoclimab in participants with CIDP who have completed Study IMVT-1401-2401 (NCT05581199). In this study, participants will receive 340 mg of batoclimab subcutaneously (SC) once weekly (QW) for up to 52 weeks. Upon completion of the Week 52 or early termination (ET) Visit, participants will transition into the 4-week Follow-up Period, which concludes with a Follow-up Visit approximately 28 (± 7) days after the Week 52 or ET Visit.

ELIGIBILITY:
Inclusion Criteria:

* Any participant who has completed Study IMVT-1401-2401
* Female participants of childbearing potential must agree to use a highly effective method of birth control
* Female participants must agree not to donate eggs throughout the study and for 90 days after the final study treatment administration
* Male participants must agree to use 1 highly effective contraception method with partners of childbearing potential throughout the study period and for 90 days after the final study treatment administration
* Male participants must agree not to donate sperm throughout the study period and for 90 days after the final study treatment administration
* Agree not to participate in another interventional study while on treatment

Exclusion Criteria:

* Participant has any medical condition (acute or chronic illness) or psychiatric condition, including autoimmune disease or neurologic disease other than CIDP, or known history of drug or alcohol abuse that, in the opinion of the Investigator, could jeopardize the participant's ability to participate in this study, compromise accurate assessment of CIDP symptoms or otherwise interfere with the course and conduct of the study.
* Participant intends to have a live vaccination during the course of the study or within 7 weeks following the final dose of batoclimab
* Participant has an ongoing SAE or a medical condition in the IMVT-1401-2401 study that the Investigator considers putting the participant at a significantly increased risk of participating in Study IMVT-1401-2402
* Participant has received Standard of Care therapy for treatment of a relapse in Study IMVT-1401-2401

Note: Other protocol specified criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants with Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and TEAEs Leading to Treatment Discontinuation | Up to 52 weeks

SECONDARY OUTCOMES:
Change from Baseline in Adjusted inflammatory Neuropathy Cause and Treatment (aINCAT) | Up to 52 weeks
  The INCAT disability scale is a widely used and validated efficacy assessment of neurologic dysfunction in CIDP and will be used for measurement of clinical response.
Change from Baseline in Mean Grip Strength | Up to 52 weeks
  Mean Grip strength provides an objective, quantitative and immediate assessment of strength impairment.

CONTACTS AND LOCATIONS:
Locations (30):
- United States (5):
  - Site Number - 1621, New Haven, Connecticut
  - Site Number - 1617, Ormond Beach, Florida
  - Site Number - 1611, Nicholasville, Kentucky
  - Site Number - 1610, Charlotte, North Carolina
  - Site Number - 1601, Austin, Texas
- Argentina (4):
  - Site Number - 7753, Rosario, Santa Fe Province
  - Site Number - 7751, Rosario, Santa Fe Province
  - Site Number - 7750, Buenos Aires
  - Site Number - 7752, San Miguel de Tucumán
- Site Number - 4680, Leuven, Vlaams Brabant, Belgium
- Brazil (3):
  - Site Number - 9103, Brasília, Federal District
  - Site Number - 9101, Curitiba, Paraná
  - Site Number - 9100, Ribeirão Preto, São Paulo
- Site Number - 6702, Leipzig, Saxony, Germany
- Greece (3):
  - Site Number - 6341, Pátrai, Achaïa
  - Site Number - 6344, Athens, Attica
  - Site Number - 6347, Larissa
- Italy (3):
  - Site Number - 6305, Bologna, Emilia-Romagna
  - Site Number - 6309, Rome, Lazio
  - Site Number - 6307, Milan, Lombardy
- Poland (6):
  - Site Number - 3207, Poznan, Greater Poland Voivodeship
  - Site Number - 3208, Krakow, Lesser Poland Voivodeship
  - Site Number - 3209, Krakow, Lesser Poland Voivodeship
  - Site Number - 3210, Lublin, Lublin Voivodeship
  - Site Number - 3206, Lublin, Lublin Voivodeship
  - Site Number - 3201, Katowice, Silesian Voivodeship
- Romania (2):
  - Site Number - 8403, Timișoara, Timiș County
  - Site Number - 8400, Constanța
- Site Number - 8501, Belgrade, Serbia
- Site Number - 8603, Prešov, Slovakia

IPD SHARING:
Plan to Share IPD: No